CLINICAL TRIAL: NCT05446077
Title: Quantitatively Analysis of Fundus Structure Characteristics in Glaucoma Following Congenital Cataract Surgery (GFCS) Using Optical Coherence Tomography Angiography
Brief Title: Quantitatively Analysis of Fundus Structure Characteristics in Glaucoma Following Congenital Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: CCMPOH2022-01
Record Dates: First submitted 2022-06-26; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Glaucoma Secondary; Congenital Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To quantitatively analyze the fundus structure and microvascular characteristics of GFCS and non-GFCS (NGFCS) using optical coherence tomography angiography (OCTA), to explore the vascular-structural association, and to assess the diagnostic abilities of structure parameters.

DETAILED DESCRIPTION:
A cross-sectional study. A total of 129 congenital cataract patients after congenital cataract extraction (40 in GFCS and 89 in NGFCS) were enrolled in this study from December 2020 to March 2021. All participants, age range from 4 to 18 years old, completed OCT examinations (including macular structure parameters, optic nerve fiber layer thickness periphery retinal nerve fiber layer [pRNFL], and sub foveal choroidal thickness [SFCT]). All the NGFCS participants underwent OCTA examinations (including vessel density (VD) and perfusion density (PD) of macular and peripapillary area.). Linear regression models were used to examine the effect of various factors on different ocular parameters. Vascular-structural associations were assessed with Spearman correlation. Diagnostic ability was evaluated with area under the receiver operating curve (AUC).

ELIGIBILITY:
NGFCS Group Inclusion Criteria:

* 1) The guardian of the child voluntarily signed the informed consent;
* 2) 4 years old ≤ age ≤ 18 years old, regardless of gender;
* 3) In line with the diagnostic criteria of NGFCS; that is, cataract extraction surgery was performed in our hospital, with no restrictions on the eye of the surgery, and implantation / or no intraocular lens implantation;
* 4) No other serious postoperative complications other than GFCS occurred after cataract extraction, such as retinal detachment, vitreous hemorrhage, choroidal detachment, etc.
* 5) The children included in this study need to have good gaze ability. Considering that the visual acuity of CC children after cataract extraction is lower than that of normal children of the same age, the best-corrected visual acuity of the included patients is ≤0.4logMAR (implanted IOL or wearing frame glasses, Contact lenses to correct vision), can better cooperate to complete OCT and OCTA examinations;

GFCS Group Inclusion Criteria:

* 1) The guardian of the child voluntarily signed the informed consent;
* 2) Clinical diagnosis of GFCS
* 3) The age of 4 years old is less than or equal to 18 years old, and the gender is not limited;
* 4) The diagnostic criteria of GFCS are met; one or both eyes are affected; Tremor, best corrected visual acuity ≤0.7logMAR, can better cooperate with OCT and OCTA examination;

The diagnostic criteria of GFCS： Childhood: based on national criteria, <18 years old (USA); 16 years old (UK, Europe,UNICEF) Childhood glaucoma: two or more of the following are required

1. Intraocular pressure: >21 mmHg (investigator discretion on method of measurement and if EUA data alone is sufficient).
2. Visual fields: reproducible visual field defect that is consistent with glaucomatous optic neuropathy with no other observable reason for the visual field defect.
3. Axial length: progressive myopia or myopic shift with increased ocular dimensions that outpace normal growth.
4. Cornea: findings including Haab striae, corneal diameter >11mm in newborns, >12mm in children younger than 1 year old, and >13mm in children older than 1 year old.
5. Optic nerve: progressive increase in cup-disc ratio, cup-disc asymmetry of 0.2 when optic discs are of similar size, and focal rim thinning.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study is a cross-sectional clinical study. Including children who were followed up in the pediatric cataract clinic of our hospital from December 1, 2020, to March 31, 2021, and had been diagnosed with GFCS, as well as patients diagnosed with non-congenital cataract extraction after surgery(NGFCS).
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Linear regression models were used to examine the effect of various factors on different ocular parameters with demographic factors. （RNFL thickness with gender, age, axial length） | December 1st 2020 to March 31st 2021
  All participants completed OCT examinations (including macular structure parameters, optic nerve fiber layer thickness periphery retinal nerve fiber layer [pRNFL], and sub foveal choroidal thickness [SFCT]). All the NGFCS participants underwent OCTA examinations (including vessel density (VD) and perfusion density (PD) of macular and peripapillary area.). Linear regression models were used to examine the effect of various factors on different ocular parameters with demographic factors.
Vascular-structural associations were assessed with Spearman correlation. (RNFL thickness and ONH vessels density, perfusion density) | December 1st 2020 to March 31st 2021
  All participants completed OCT examinations (including macular structure parameters, optic nerve fiber layer thickness periphery retinal nerve fiber layer [pRNFL], and sub foveal choroidal thickness [SFCT]). All the NGFCS participants underwent OCTA examinations (including vessel density (VD) and perfusion density (PD) of macular and peripapillary area.). Vascular-structural associations were assessed with Spearman correlation.
Diagnostic ability of GFCS was evaluated with area under the receiver operating curve (AUC). | December 1st 2020 to March 31st 2021
  All participants completed OCT examinations (including macular structure parameters, optic nerve fiber layer thickness periphery retinal nerve fiber layer [pRNFL], and sub foveal choroidal thickness [SFCT]). All the NGFCS participants underwent OCTA examinations (including vessel density (VD) and perfusion density (PD) of macular and peripapillary area.). Diagnostic ability of GFCS was evaluated with area under the receiver operating curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China